CLINICAL TRIAL: NCT04951635
Title: A Phase III, Randomised, Double-blind, Placebo-controlled, Multi-centre Study of Almonertinib as Maintenance Therapy in Patients With Locally Advanced, Unresectable EGFR Mutation-positive Non-Small Cell Lung Cancer (Stage III) Who Have Not Progressed Following Definitive, Platinum-based Chemoradiation Therapy
Brief Title: A Phase III Study to Assess the Effects of Almonertinib Following Chemoradiation in Patients With Stage III Unresectable Non-small Cell Lung Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HS-10296-304
Record Dates: First submitted 2021-06-30; First posted 2021-07-07 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Phase III, stage III NSCLC, unresectable NSCLC, Almonertinib, Maintenance Therapy, EGFR, chemoradiation therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — aumolertinib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Almonertinib (Experimental)
  Interventions: Drug: Almonertinib
- Placebo Almonertinib (Placebo Comparator)
  Interventions: Drug: Placebo Almonertinib

INTERVENTIONS:
Drug: Almonertinib — The initial dose of Almonertinib 110 mg daily can be reduced to 55 mg daily under specific conditions.
  Treatment can continue until disease progression, unacceptable toxicity or other discontinuation criteria are met. The 2:1 ratio (Almonertinib to placebo).
  Other Names: HS-10296
  Arms: Almonertinib
Drug: Placebo Almonertinib — The initial dose of Placebo Almonertinib 110 mg daily can be reduced to 55 mg daily under specific conditions.
  Treatment can continue until disease progression, unacceptable toxicity or other discontinuation criteria are met. The 2:1 ratio (Almonertinib to placebo).
  Arms: Placebo Almonertinib

SUMMARY:
To assess the efficacy and safety of Almonertinib versus placebo following chemoradiation in patients with stage III unresectable epidermal growth factor receptor mutation-positive (EGFRm+) non-small cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, multicenter, phase III study to assess the efficacy and safety of Almonertinib following chemoradiation in patients with stage III unresectable EGFRm+ NSCLC, including the most common EGFR sensitizing mutations (Ex19Del and L858R), either alone or in combination with other EGFR mutations (e.g., T790M). Chemoradiation may have been given either concurrently or sequentially. Patients whose disease has not progressed following chemoradiation will be randomised within 6 weeks of completion of chemoradiation to receive Almonertinib or placebo in a 2:1 ratio, and treatment will be continued until disease progression, unacceptable toxicity or other discontinuation criteria are met. After progression, patients can be unblinded and may receive open-label Almonertinib for as long as their treating physician considers they are deriving clinical benefit.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent before any study-specific procedures, sampling and analyses.
2. Male or female, age at least 18 years.
3. Histologically or cytologically confirmed diagnosis of primary non-small lung cancer (NSCLC) on predominantly non-squamous pathology who present with locally advanced, unresectable (Stage III) disease (according to AJCC 8th edition lung cancer classification). Recommended by not required: In addition to obvious cT4 disease, lymph node status N2 or N3 should be confirmed by intrabronchial ultrasound, mediastinoscopy or thoracoscopy biopsy, and under the condition of no biopsy or negative biopsy, the whole body screening of 18F-Fluro-deoxyglucose positron emission tomography (PET)or contrast agent-enhanced computed tomography (CT) to confirm.
4. The tumor harbours one of the two common EGFR mutations known to be associated with EGFR-TKI sensitivity (Ex19Del, L858R), either alone or in combination with other EGFR mutations including T790M, assessed by cobas® EGFR Mutation Test (Roche Diagnostics) or Xiamen AmoyDx EGFR (ADx-ARMS, Super-ARMS method) kit in site or central laboratory.
5. Patients must have received either concurrent chemoradiation or sequential chemoradiation including at least 2 cycles of platinum based chemotherapy and a total dose of radiation of 60 Gy ±10% (54 to 66 Gy).
6. Chemoradiation must be completed ≤6 weeks prior to randomization.
7. Patients must not have had disease progression during or following definitive platinum-based, chemoradiation therapy.
8. A WHO performance status of 0-1 with no deterioration over the past 2 weeks and a minimum life expectancy of 12 weeks.
9. Female patients should be using adequate contraceptive measures and should not be breastfeeding at the screening period, during the study, and six months after the last dosing of study. A pregnancy test should be done before first dosing unless having evidence of non-child-bearing potential.
10. Male patients should be willing to use barrier contraception (condoms)

Exclusion Criteria:

1. Treatment with any of the following:

   1. Prior treatment with any prior chemotherapy, radiation therapy, immunotherapy or investigational agents for NSCLC outside of that received in the definitive setting for Stage III disease (chemotherapy and radiotherapy in SCRT and CCRT regimens is allowed for treatment of Stage III disease). Patients who have previously undergone surgery for stage I or stage II NSCLC can be enrolled. If neoadjuvant or adjuvant therapy (non-EGFR tyrosine kinase inhibitor) is used, neoadjuvant or adjuvant therapy needs to be completed for at least half a year (6 months) before enrollment.
   2. Prior treatment with EGFR-TKI therapy.
   3. Major surgery (including primary tumor surgery, excluding placement of vascular access) within 4 weeks of the first dose of study drug.
   4. Patients currently receiving (unable to stop use prior to receiving the first dose of study treatment) medications or herbal supplements known to be strong inducers and inhibitors of cytochrome CYP3A4 (at least 7 days prior to receiving the first dose of study drug).
   5. Treatment with an investigational drug within five half-lives of the compound or any of its related material.
2. Mixed small cell and non-small cell lung cancer histology.
3. History of interstitial lung disease (ILD) prior to chemoradiation.
4. Symptomatic pneumonitis following chemoradiation.
5. Inadequate bone marrow reserve or organ function.
6. Any unresolved toxicity Common Terminology Criteria for Adverse Events (CTCAE) ≥ Grade 2 from the prior chemoradiation therapy.
7. Any of the following cardiac criteria:

   1. Mean resting corrected QT interval (QTc) > 470 ms obtained from 3 electrocardiograms (ECGs), using the screening clinic's ECG machine and Fridericia's formula for QT interval correction (QTcF).
   2. Any clinically important abnormalities in rhythm, conduction, or morphology of the resting ECG (e.g., PR interval > 250 ms).
   3. Any factors that increase the risk of QTc prolongation or risk of arrhythmic events, such as heart failure or any concomitant medication known to prolong the QT interval.
   4. Left ventricular ejection fraction (LVEF) ≤ 40%.
8. History of other malignancies, excluding fully treated non-melanoma skin cancer, in-situ cancer, or other solid tumors that hadn't recurrent for > 5 years following the end of treatment.
9. Any evidence of severe or uncontrolled systemic diseases (including uncontrolled hypertension and active bleeding diatheses) or active infection (including hepatitis B, hepatitis C, and human immunodeficiency virus (HIV)).
10. Refractory nausea, vomiting, or chronic gastrointestinal diseases, or inability to swallow the study drug that would preclude adequate absorption of Almonertinib.
11. History of hypersensitivity to any active or inactive ingredient of Almonertinib or to drugs with a similar chemical structure or class to Almonertinib.
12. Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions, and requirements.
13. Any severe and uncontrolled ocular disease that may, in the ophthalmologist's opinion, present a specific risk to the patient's safety.
14. Any disease or condition that, in the opinion of the investigator, would compromise the safety of the patient or interfere with study assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-03-18 (Actual); Primary Completion 2024-07-15 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) assessed by IRC (Independent Review Committee) | Tumor scans performed at baseline then every ~8 weeks up to 48 weeks, then every ~12 weeks thereafter until confirmed disease progression; up to a maximum of approximately 3 years.
  Progression-free survival (PFS) assessed by IRC (Independent Review Committee) Description: PFS is defined as the time from randomization until the date of objective disease progression or death (by any cause in the absence of progression) regardless of whether the patient withdraws from randomised therapy or receives another anti-cancer therapy prior to progression, based on blinded independent central review assessment according to RECIST 1.1.

SECONDARY OUTCOMES:
PFS assessed by INVs (Investigators) | Tumor scans performed at baseline then every ~8 weeks up to 48 weeks, then every ~12 weeks thereafter until confirmed disease progression; up to a maximum of approximately 3 years.
  PFS is defined as the time from randomization to progression of tumor as assessed by INVs or death from any cause on study.
Time to CNS PFS assessed by IRC | Tumor scans performed at baseline then every ~8 weeks up to 48 weeks, then every ~12 weeks thereafter until confirmed disease progression; up to a maximum of approximately 3 years.
  Defined as earlier event of CNS progression or death based on blinded independent central review assessment according to RECIST 1.1.
Overall survival (OS) | From baseline until death due to any cause; up to a maximum of approximately 4 years.
  OS is deﬁned as the time from the date of randomization until death due to any cause.
Objective response rate (ORR) | Tumor scans performed at baseline then every ~8 weeks up to 48 weeks, then every ~12 weeks thereafter until confirmed disease progression; up to a maximum of approximately 4 years.
  Defined as the number (%) of patients with measurable disease with at least 1 visit response of CR (Complete response) or PR (Partial response) based on blinded independent central review assessment according to RECIST 1.1.
Duration of response (DoR) | Tumor scans performed at baseline then every ~8 weeks up to 48 weeks, then every ~12 weeks thereafter until confirmed disease progression; up to a maximum of approximately 4 years.
  Defined as the time from the date of first documented response (i.e., subsequently confirmed) until the date of documented progression or death in the absence of disease progression based on blinded independent central review assessment according to RECIST 1.1.
Disease control rate (DCR) | Tumor scans performed at baseline then every ~8 weeks up to 48 weeks, then every ~12 weeks thereafter until confirmed disease progression; up to a maximum of approximately 4 years.
  Defined as Disease control rate is defined as the percentage of subjects who have a best overall response of CR or PR or SD based on blinded independent central review assessment according to RECIST 1.1.
Time to death or distant metastases (TTDM) | Tumor scans performed at baseline then every ~8 weeks up to 48 weeks, then every ~12 weeks thereafter until confirmed disease progression; up to a maximum of approximately 4 years.
  Defined as the time from the date of randomization until the first date of distant metastasis or date of death in the absence of distant metastasis based on blinded independent central review assessment according to RECIST 1.1
Incidence of Adverse Events (AEs) | From the screening period to 28 days after treatment completion, approximately 4 years.
  AEs are graded according to CTCAE v5.0 and recorded in the case report form.

CONTACTS AND LOCATIONS:
Locations (1):
- Shandong Cancer Hospital, Ji'nan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided